CLINICAL TRIAL: NCT06370182
Title: A Prospective, Randomized, Dual-arm Multi-center Study to Assess the Safety and Effectiveness of Mechanical Thrombectomy Using the Anaconda ANA Funnel Catheter in Combination With a Stent Retriever
Brief Title: Safety and Effectiveness of Mechanical Thrombectomy Using the Anaconda ANA Funnel Catheter
Acronym: ATHENA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anaconda Biomed S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANA2401
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: flow arrest; flow restriction; funnel; guide catheter; mechanical thrombectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ANA Funnel Catheter Group (Experimental): Mechanical thrombectomy using a stent retriever delivered by the ANA device.
  Interventions: Device: ANA Funnel Catheter
- Control Group (Active Comparator): Mechanical thrombectomy using a stent retriever delivered by an approved guide catheter.
  Interventions: Device: Control

INTERVENTIONS:
Device: ANA Funnel Catheter — Mechanical thrombectomy using a stent retriever delivered by the ANA device that enables local flow restriction when deployed.
  Arms: ANA Funnel Catheter Group
Device: Control — Mechanical thrombectomy using a stent retriever delivered by an approved guide catheter with or without an intermediate catheter and aspiration per conventional techniques.
  Arms: Control Group

SUMMARY:
The objective of this study is to assess the safety and effectiveness of mechanical thrombectomy (MT) using the ANA funnel catheter in its intended use, which is to facilitate the navigation and deployment of other neurovascular devices and to allow flow arrest during mechanical thrombectomy procedures performed in subjects experiencing acute ischemic stroke (AIS) secondary to large vessel occlusion (LVO) and treated within 24 hours of symptom onset.

DETAILED DESCRIPTION:
Similar to other ancillary devices used in MT, the ANA device is designed to facilitate the delivery of stent retrievers and other catheters during these procedures. Its design aims to enhance procedural success and the efficiency of stent retriever-based MT by enabling flow arrest during clot retrieval. This approach has been shown to improve rates of revascularization and favorable clinical outcomes at three months.

The use of the ANA to facilitate MT with a stent retriever may provide a simplified approach to flow restriction and could achieve acute reperfusion outcomes comparable to commonly used strategies that combine direct aspiration with an intermediate catheter to actuate clot retrieval with a SR.

A dual-arm, prospective, randomized study will be conducted to demonstrate the safety and effectiveness of ANA compared to a conventional approach using cleared stent retrievers for MT. The study will report acute reperfusion success after a single thrombectomy pass with three of the most commonly employed stent retrievers: Solitaire, Trevo, and pRESET. Procedural safety will be assessed by comparing the rate of procedure-related sICH within 24 hours of the intervention between study arms.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects meeting all inclusion criteria will be considered for enrollment in the study.

1. Age 22 to 85 years.
2. Informed consent was obtained from subject or acceptable subject surrogate (e.g., next of kin, or legal representative).
3. A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
4. Baseline NIHSS obtained prior to procedure ≥ 6 points and ≤ 25 points.
5. Pre-ictal mRS score of 0,1 or 2.
6. Treatable within 16 hours of symptom onset, defined as point in time when the subject was last observed to be asymptomatic; treatment start is defined by arterial puncture time.
7. If indicated, thrombolytic therapy shall be initiated per the institution's usual care and the most recent version of the AHA/ASA Guidelines. Subjects eligible for IV thrombolysis should receive it without delay.
8. Occlusion (eTICI ≤ 1 flow) of the terminal carotid artery, middle cerebral artery M1 segment or, dominant or proximal M2 segment, indicated for mechanical thrombectomy, confirmed with conventional angiography or CTA/MRA.
9. Imaging criteria:

   * Perfusion weighted criterion: volume of diffusion restriction visually assessed

     ≤ 50 mL on CTP/MRP, or
   * CT criterion: Alberta Stroke program early CT score (ASPECTS) 6 to 10 on baseline CT/DWI-MRI. (Inclusion of subjects with ASPECTS 5 is permitted at centers performing scoring on MRI)
10. The subject is indicated for a neurovascular thrombectomy procedure with an approved stent retriever per its Instructions for Use.

Key Exclusion Criteria:

Subjects who meet any of the exclusion criteria will be ineligible for participation in the study.

The following exclusion criteria will be assessed pre-operatively:

1. Subject was diagnosed with a stroke in the past year.
2. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
3. Known hemorrhagic diathesis, coagulation factor deficiency, oral anticoagulant therapy with antivitamin K, with INR >3.0, or thrombocytopenia - baseline platelet count < 50,000 platelets/mL.
4. Known baseline glucose of <50 mg/dL or >400 mg/dL.
5. Severe, sustained uncontrolled hypertension refractory to treatment (systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg).
6. Serious, advanced, or terminal disease with anticipated life expectancy of less than 1 year.
7. Known cancer with metastases.
8. History of life-threatening allergy (more than rash) to contrast medium.
9. Known renal insufficiency with creatinine ≥3 mg/dL or glomerular filtration rate (GFR) <30 mL/min.
10. Subject is a current user or has a recent history of cocaine &/or heroin use.
11. Known pregnancy and/or lactating female.
12. Subject is participating in a concurrent study involving an investigational drug or device that would impact the primary endpoint of this study.
13. Subject is unlikely to be available for a 90-day follow-up (e.g. no fixed home address, visitor from overseas, etc.)
14. CT or MRI evidence of hemorrhage (the presence of microbleeds is allowed).
15. Significant mass effect with midline shift.
16. Evidence of intracranial tumor (except asymptomatic meningioma of ≤ 2cm in diameter).
17. Suspicion of aortic dissection, presumed septic embolus, or suspicion of bacterial endocarditis.
18. History of preexisting stent proximal to or at the occlusion site that may preclude safe deployment or recovery of the stent retriever.
19. Vessel tortuosity too difficult to allow endovascular access of the intracranial ICA per investigator judgement. Indicators of vessel tortuosity include but are not limited to the presence of carotid loops and type 3 aortic arches.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with "near-complete" reperfusion after one thrombectomy pass (FPE, eTICI 2c-3, extended Thrombolysis in Cerebral Infarction scale) in the target vessel. | intra-operative
  Reperfusion (eTICI 2c-3) to be assessed by an independent Core Lab.
Rate of symptomatic intracranial hemorrhage (sICH), attributable to the device or procedure. | Within 24 hours of the procedure
  Extent of hemorrhage to be assessed by an independent Core Lab, symptoms to be assessed by the Data Monitoring Committee (DMC).

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Siddiqui, MD, PhD, FAHA, Principal Investigator — Jacobs School of Medicine & Biomedical Sciences; Santiago Ortega-Gutierrez, MD, MSc, FAHA, FSVIN, Principal Investigator — University of Iowa
Locations (22):
- United States (11):
  - Baptist Health Medical Center, Jacksonville, Florida
  - Grady Memorial Hospital, Emory, Atlanta, Georgia
  - Advocate Health, Park Ridge, Illinois
  - University of Iowa, Iowa City, Iowa
  - Boston Medical Center, Boston, Massachusetts
  - University of Buffalo Neurosurgery, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- France (4):
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Fondation Rothschild, Paris
  - Hospital Foch, Suresnes
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Semmelweis University Hospital, Budapest, Hungary
- Spain (5):
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
- Aydin University Hospital, Istanbul, Turkey (Türkiye)